CLINICAL TRIAL: NCT05645055
Title: The Clinical Outcomes of Patients With Stricturing Crohn's Diseases Received Biologics: a Prospective, Observative Study
Brief Title: Biologics for Stricturing Crohn's Diseases
Status: Recruiting | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Weiming, Senior Doctor, Principal Investigator, Clinical Professor, Jinling Hospital, China
Other Study IDs: JinlingH20221203
Record Dates: First submitted 2022-12-02; First posted 2022-12-09 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: The Efficacy of Biologics for Stricturing Crohn's Diseases
MeSH Terms: interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with stricturing Crohn's diseases: Patients with stricturing Crohn's diseases
  Interventions: Other: treat these patients with biologics

INTERVENTIONS:
Other: treat these patients with biologics — treat these patients with biologics

SUMMARY:
Recent researches have reported that biologics might be also effective for stricturing CD. However, the data were largely retrospective. Prospective studied are needed for evaluate the efficacy of biologics for stricturing Crohn's diseases.

ELIGIBILITY:
Inclusion Criteria:

* patients with stricturing Crohn's diseases
* no surgical indication
* patients with asymptomatic penetrating diseases
* written consent acquired

Exclusion Criteria:

* patients with surgical indication
* patients with symptomatic penetrating diseases
* contraindication of biologics
* anticipating other trial

Ages: 16 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 200
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
clinical remission rate at 1 year | clinical remission rate at 1 year
  clinical remission rate at 1 year (CDAI less than 150)

SECONDARY OUTCOMES:
clinical remission rate at 5 year | clinical remission rate at 5 year
  clinical remission rate at 5 year (CDAI less than 150)
surgical recurrence rate at 1 and 5 year | at 1 and 5 year
  surgical recurrence : needing surgery for CD recurrence
endoscopic recurrence rate at 1 and 5 year | at 1 and 5 year
  endoscopic recurrence: rutgeerts over i2b
quality of life of patients assessed by IBDQ | at 2, 4, 6 , 8 months and at 1, 2, 3, 4 and 5 year
  IBDQ
quality of life of patients assessed by Short form 12 | at 2, 4, 6 , 8 months and at 1, 2, 3, 4 and 5 year
  Short form 12
score of obstructive | at 2, 4, 6 , 8 months and at 1, 2, 3, 4 and 5 year
  range 0-6, higher means severe

CONTACTS AND LOCATIONS:
Overall Officials: Weiming wm Zhu, Ph.D., Principal Investigator — Jinling Hospital, China
Locations (1):
- Department of General Surgery, Jinling hosptal,Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided